CLINICAL TRIAL: NCT05981612
Title: Effects of Emotional Reactivity on Decision-Making in Adolescents With Nonsuicidal Self-Injury
Brief Title: Impact of Emotional Reactivity on Dysfunctional Decision-Making in NSSI Adolescents
Status: Recruiting | Type: Observational
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Other Study IDs: BAM_lab_NSSI_04
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nonsuicidal Self Injury; Prediction Errors
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSSI
- HC

SUMMARY:
Nonsuicidal self-injury (NSSI) is defined as direct, intentional physical injury without suicidal intention. Studies revealed that dysfunctional interpersonal relationships and reward-related decision-making may play crucial roles in this maladaptive behavior, especially in adolescents. These interpersonal decision contexts are characterized by constant updating of expectations of rewards and the actual received rewards as well as the associated emotional reactions. These processes have recently been computationally formalized as prediction errors (PE), specifically reward PEs, valence PEs, and arousal PEs (Heffner et al., 2021; Nat Hum Behav). In the current study, the investigators aim to investigate whether these PEs make discernible contributions to social decisions in the context of unfair experiences among adolescents with NSSI and matched healthy control adolescents (HC). Specifically the investigators hypothesized that: 1) reward and emotional PEs show significant predictions of punishment decisions in both groups, 2) however, compared to HC adolescents, the NSSI group will exhibit selective dysfunctions in emotional but not reward PEs leading to punish a norm proposer who provided unfair offers.

ELIGIBILITY:
Inclusion Criteria:

* 15-18 years
* right-handed
* normal or corrected normal visual acuity
* meet the proposed DSM-5 frequency criteria (e.g., ≥5 days of NSSI behaviors in the past year)

Exclusion Criteria:

* diagnosis of borderline personality disorder, major depressive disorder, other
* psychiatric disorders, etc.
* high suicidal risk
* recent use of medications that can affect neural activity
* have received or are receiving Dialectical Behavior Therapy (DBT) other treatment for emotional problems within the past 6 months
* have a contraindication to MRI scanning (e.g., metal implants, claustrophobia or other conditions that make them inappropriate for MRI scanning)

Ages: 15 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Treatment-seeking NSSI individuals will be recruited from local hospitals and HC from the community.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Reward prediction errors (PEs) | About 20 minutes
  Reward PEs will be calculated by the differences between the experienced (when be offered) reward and predicted (before the offer) reward.
Valence prediction errors (PEs) | About 20 minutes
  Valence PEs will be calculated by the differences between the experienced emotional valence and predicted emotional valence.
Arousal prediction errors (PEs) | About 20 minutes
  Arousal PEs will be calculated by the differences between the experienced emotional arousal and predicted emotional arousal.
The prediction of PEs of punishment decisions | About 20 minutes
  All PEs and groups (NSSI, HC) will be used in a regression model to examined whether there is any alteration in the NSSI group when PEs are predicted to punishment (reject) decisions.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial Center for Mental Health, Sichuan Provincial People's Hospital, University of Electronic Science and Technology of China, Chengdu, Sichuan, China